CLINICAL TRIAL: NCT02155660
Title: A Randomised, Double-blind, Double Dummy, 56 Week Placebo-controlled, Multicentre, Parallel Group, Phase 3 Study Evaluating Efficacy/Safety of 3 Benralizumab Doses in Patients With Moderate to Very Severe COPD With Previous Exacerbations.
Brief Title: Efficacy and Safety of Benralizumab in Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD) With Exacerbation History
Acronym: TERRANOVA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3251C00004
Record Dates: First submitted 2014-05-20; First posted 2014-06-04 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Keywords: Obstructive Lung Diseases; Chronic Obstructive Pulmonary Disease; Lung Disease; Bronchial Diseases; COPD Exacerbation; Respiratory Tract Diseases
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive; Lung Diseases; Bronchial Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Benralizumab Arm A (Experimental): Benralizumab administered subcutaneously
  Interventions: Drug: Benralizumab Arm A
- Benralizumab Arm B (Experimental): Benralizumab administered subcutaneously
  Interventions: Drug: Benralizumab Arm B
- Benralizumab Arm C (Experimental): Benralizumab administered subcutaneously
  Interventions: Drug: Benralizumab Arm C
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benralizumab Arm A — Benralizumab subcutaneously on study week 0 until study week 48 inclusive
  Arms: Benralizumab Arm A
Drug: Benralizumab Arm B — Benralizumab subcutaneously on study week 0 until study week 48 inclusive
  Arms: Benralizumab Arm B
Drug: Benralizumab Arm C — Benralizumab subcutaneously on study week 0 until study week 48 inclusive
  Arms: Benralizumab Arm C
Drug: Placebo — Benralizumab subcutaneously on study week 0 until study week 48 inclusive
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if benralizumab reduces COPD exacerbation rate in symptomatic patients with moderate to very severe COPD who are receiving standard of care therapies.

ELIGIBILITY:
Inclusion Criteria:.

* Informed consent.
* Subjects 40-85 y.o.
* Moderate to very severe COPD with Post Bronchodilator (BD) FEV1>20% and ≤65%.

  -≥2 moderate or ≥1 severe COPD exacerbation(s) required treatment or hospitalization within 2-52 weeks prior to Visit1.
* Modified Medical Research Council (mMRC) score ≥1 at Visit 1.
* Treatment with double or triple therapy throughout the year prior to Visit 1, constant 2 weeks prior to Visit 1.
* Tobacco history of ≥10 pack-years.
* Women of childbearing potential must use a highly effective form of birth control from Visit 1 until 16 weeks after their last dose, and negative serum pregnancy test result at Visit 1.
* Male subjects who are sexually active must be surgically sterile one year prior to Visit 1 or use an adequate method of contraception from the first Investigational Product (IP) dose until 16 weeks after their last dose.
* Compliance with maintenance therapy during run-in ≥70%.
* Blood eosinophils due to subject's stratification and cap for blood eosinophil levels.When any eosinophil cohort is full, subjects in the completed cohort will not be randomised and will be withdrawn from the study.

Exclusion criteria:

* Clinically important pulmonary disease other than COPD or another diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts.
* Any disorder or major physical impairment that is not stable by Investigator opinion and/or could affect: - subject safety-study findings or their interpretation or subject's ability to complete the entire study duration.
* Unstable ischemic heart disease, arrhythmia, cardiomyopathy, or other relevant cardiovascular disorder that in Investigator's judgment may put the patient at risk or negatively affect the study outcome.
* Treatment with systemic corticosteroids and/or antibiotics, and/or hospitalization for a COPD exacerbation within 2 weeks prior to Visit1 or during the enrolment and run-in period.
* Acute upper or lower respiratory infection requiring antibiotics within 2 weeks prior to Visit1 or during the enrolment and run-in period.
* Pneumonia within 8 weeks prior to Visit1 or during the enrolment and run-in period.
* Pregnant, breastfeeding, or lactating women.
* Risk factors for pneumonia
* History of anaphylaxis to any other biologic therapy.
* Long term oxygen therapy with signs and/or symptoms of cor pulmonale, right ventricular failure.
* Use of immunosuppressive medication within 2 weeks prior to Visit1 and/or during the enrolment and run-in period.
* Receipt of any investigational non-biologic product within 30 days or 5 half-lives prior to Visit 1.
* Evidence of active tuberculosis (TB) without an appropriate course of treatment.
* Lung volume reduction surgery within the 6 months prior to Visit 1. History of partial or total lung resection (single lobe or segmentectomy is acceptable).
* Asthma as a primary or main diagnosis according to the Global Initiative for Asthma (GINA) guidelines or other accepted guidelines.
* Previous treatment with benralizumab.
* Helminth parasitic infection diagnosed within 24 weeks prior to Visit 1.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2255 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bartolome R. Celli, MD, Principal Investigator — Brigham and Women's Hospital, Pulmonary Division, 75 Francis Street, PBB Clinics 3, Boston, MA 02115
Locations (293):
- United States (130):
  - Research Site, Birmingham, Alabama
  - Research Site, Gulf Shores, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Flagstaff, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Anaheim, California
  - Research Site, Arcadia, California
  - Research Site, Bakersfield, California
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, Hawaiian Gardens, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Palmdale, California
  - Research Site, Peninsula, California
  - Research Site, Placentia, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Westminster, California
  - Research Site, Centennial, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Chiefland, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coconut Creek, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, DeBary, Florida
  - Research Site, DeLand, Florida
  - Research Site, Doral, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Miami, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sarasota, Florida
  - Research Site, South Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Nampa, Idaho
  - Research Site, Evergreen Park, Illinois
  - Research Site, O'Fallon, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, River Forest, Illinois
  - Research Site, Topeka, Kansas
  - Research Site, Henderson, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Opelousas, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Sunset, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Lutherville, Maryland
  - Research Site, White Marsh, Maryland
  - Research Site, Fall River, Massachusetts
  - Research Site, Marlborough, Massachusetts
  - Research Site, Buckley, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Fridley, Minnesota
  - Research Site, Woodbury, Minnesota
  - Research Site, Picayune, Mississippi
  - Research Site, Port Gibson, Mississippi
  - Research Site, Belton, Missouri
  - Research Site, Florissant, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Fremont, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Marlton, New Jersey
  - Research Site, Union, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Great Neck, New York
  - Research Site, Mineola, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Potsdam, New York
  - Research Site, The Bronx, New York
  - Research Site, Burlington, North Carolina
  - Research Site, Calabash, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Shelby, North Carolina
  - Research Site, Chardon, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Clackamas, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Monroeville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Uniontown, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Hodges, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Tullahoma, Tennessee
  - Research Site, Corsicana, Texas
  - Research Site, Dallas, Texas
  - Research Site, Duncanville, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Huntsville, Texas
  - Research Site, Killeen, Texas
  - Research Site, Lampasas, Texas
  - Research Site, Longview, Texas
  - Research Site, Lufkin, Texas
  - Research Site, McKinney, Texas
  - Research Site, Plano, Texas
  - Research Site, Sealy, Texas
  - Research Site, Bountiful, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Abingdon, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Everett, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Kingwood, West Virginia
  - Research Site, Morgantown, West Virginia
- Argentina (16):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autónoma de Buenos Aire
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Concepción del Uruguay
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Florida
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Nueve de Julio
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Fernando
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
- Australia (6):
  - Research Site, Clayton
  - Research Site, Gosford
  - Research Site, Murdoch
  - Research Site, Nedlands
  - Research Site, New Lambton
  - Research Site, Woolloongabba
- Belgium (7):
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Jambes
  - Research Site, Leuven
  - Research Site, Malmedy
  - Research Site, Turnhout
  - Research Site, Veurne
- Brazil (7):
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Sorocaba
  - Research Site, Vitória
- Bulgaria (13):
  - Research Site, Dupnitsa
  - Research Site, Kozloduy
  - Research Site, Pazardzhik
  - Research Site, Pernik
  - Research Site, Petrich
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sandanski
  - Research Site, Silistra
  - Research Site, Sofia
  - Research Site, Vidin
  - Research Site, Vratsa
  - Research Site, Yambol
- Chile (4):
  - Research Site, Curicó
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talca
- Colombia (7):
  - Research Site, Armenia
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Manizales
  - Research Site, Medellín
  - Research Site, Medillin
- Research Site, Petrinja, Croatia
- Denmark (6):
  - Research Site, Aarhus N
  - Research Site, København NV
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Roskilde
  - Research Site, Silkeborg
- France (10):
  - Research Site, Bois-Guillaume
  - Research Site, Brest
  - Research Site, La Tronche
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nîmes
  - Research Site, Orléans
  - Research Site, Pessac
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Mexico (4):
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
- New Zealand (5):
  - Research Site, Auckland
  - Research Site, Dunedin
  - Research Site, Greenlane
  - Research Site, Hamilton West
  - Research Site, Tauranga
- Norway (3):
  - Research Site, Bodø
  - Research Site, Kolbjørnsvik
  - Research Site, Svelvik
- Peru (3):
  - Research Site, Cusco
  - Research Site, Lima
  - Research Site, Piura
- Philippines (4):
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (19):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gorzów Wlkp
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Karczew
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Ostrów Wielkopolski
  - Research Site, Ruda Śląska
  - Research Site, Skierniewice
  - Research Site, Sosnowiec
  - Research Site, Starachowice
  - Research Site, Szczecin
  - Research Site, Słupca
  - Research Site, Trzebnica
  - Research Site, Wroclaw
  - Research Site, Żnin
- Research Site, Belgrade, Serbia
- Slovenia (5):
  - Research Site, Celje
  - Research Site, Golnik
  - Research Site, Kamnik
  - Research Site, Ljubljana
  - Research Site, Maribor
- Sweden (6):
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Uppsala
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (6):
  - Research Site, Bangkok
  - Research Site, Bangkoknoi
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang,
  - Research Site, Nonthaburi
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Mersin
- Ukraine (11):
  - Research Site, Cherkasy
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
- Vietnam (3):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Criner GJ, Celli BR, Singh D, Agusti A, Papi A, Jison M, Makulova N, Shih VH, Brooks L, Barker P, Martin UJ, Newbold P. Predicting response to benralizumab in chronic obstructive pulmonary disease: analyses of GALATHEA and TERRANOVA studies. Lancet Respir Med. 2020 Feb;8(2):158-170. doi: 10.1016/S2213-2600(19)30338-8. Epub 2019 Sep 28. PMID 31575508
- [Derived] Criner GJ, Celli BR, Brightling CE, Agusti A, Papi A, Singh D, Sin DD, Vogelmeier CF, Sciurba FC, Bafadhel M, Backer V, Kato M, Ramirez-Venegas A, Wei YF, Bjermer L, Shih VH, Jison M, O'Quinn S, Makulova N, Newbold P, Goldman M, Martin UJ; GALATHEA Study Investigators; TERRANOVA Study Investigators. Benralizumab for the Prevention of COPD Exacerbations. N Engl J Med. 2019 Sep 12;381(11):1023-1034. doi: 10.1056/NEJMoa1905248. Epub 2019 May 20. PMID 31112385
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2563&filename=D3251C00004%20-%20%20%20Statistical%20Analysis%20Plan_Redacted.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2563&filename=Terranova%20CSP%20and%20last%20amendment_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2255 patients signed informed consent and were randomized to received treatment with benralizumab 10 mg,30 mg, 100 mg or placebo. One participant was excluded from the analysis. Therefore results are provided for 2254 participants.
Groups:
- Benralizumab 10 mg; Benralizumab 30 mg; Benralizumab 100 mg; Placebo: Every 8 weeks administered subcutaneously
Period: Overall Study
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Started | 562 | 562 | 562 | 568
Completed | 504 | 489 | 502 | 507
Not Completed | 58 | 73 | 60 | 61
Not completed — Other Reason | 8 | 6 | 10 | 10
Not completed — Study-specific withdrawal criteria | 0 | 1 | 1 | 1
Not completed — Severe non-compliance | 0 | 4 | 0 | 1
Not completed — Adverse Event | 2 | 6 | 3 | 1
Not completed — Lost to Follow-up | 3 | 6 | 5 | 8
Not completed — Death | 17 | 19 | 17 | 19
Not completed — Withdrawal by Subject | 28 | 31 | 24 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo | Total
Number analyzed (Participants) | 562 | 562 | 562 | 568 | 2254
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Full analysis set
  Years | 64.7 (8.47) | 65.6 (8.61) | 65.0 (8.23) | 65.3 (8.44) | 65.2 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    Female | 196 | 194 | 207 | 209 | 806
    Male | 366 | 368 | 355 | 359 | 1448
Race/Ethnicity, Customized [Number; unit: participants] — Population: Full analysis set
  participants
    White | 441 | 444 | 443 | 446 | 1774
    Black or African American | 8 | 12 | 16 | 19 | 55
    Asian | 70 | 69 | 67 | 67 | 273
    Other | 43 | 37 | 36 | 36 | 152

OUTCOME MEASURES:

1. Primary Outcome: Annual COPD Exacerbation Rate Over 56 Weeks Treatment Comparison for Patients With Baseline EOS>=220/uL
Description: A COPD exacerbation is defined by symptomatic worsening of COPD requiring:
  * Use of systemic corticosteroids for at least 3 days; a single depot injectable dose of corticosteroids will be considered equivalent to a 3-day course of systemic corticosteroids; and/or
  * Use of antibiotics; and/or
  * An inpatient hospitalization or death due to COPD Annual COPD exacerbation rate is the number of exacerbations per year. Its raw rate is calculated by number of exacerbations divided by the treatment period and then normalized to an annual rate, and is estimated by negative binomial model. Rate ratio between two treatment groups is also estimated through this model.
Time Frame: Immediately following the first IP dose through week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 377 | 394 | 386 | 388
Exacerbations per year | 0.99 [0.87 to 1.13] | 1.21 [1.08 to 1.37] | 1.09 [0.96 to 1.23] | 1.17 [1.04 to 1.32]
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Test type: Superiority; p = 0.0638, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, number of exacerbations in the previous year; Rate ratio = 0.85, 95% CI 2-sided [0.71 to 1.01]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.6575, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, number of exacerbations in the previous year; Rate ratio = 1.04, 95% CI 2-sided [0.88 to 1.23]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.3988, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, number of exacerbations in the previous year; Rate ratio = 0.93, 95% CI 2-sided [0.78 to 1.10]

2. Secondary Outcome: Annual COPD Exacerbation Rate Over 56 Weeks Treatment Comparison for Patients With Baseline EOS<220/uL
Description: as for outcome 1
Time Frame: Immediately following the first IP dose through week 56
Population: Full analysis set, baseline EOS<220/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 185 | 168 | 176 | 180
Exacerbations per year | 1.23 [1.03 to 1.46] | 1.27 [1.05 to 1.53] | 1.21 [1.00 to 1.45] | 1.18 [0.98 to 1.41]
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Test type: Superiority; p = 0.7564, Negative binomial; Model includes treatment group, region, background therapy, number of exacerbations in the previous year; Rate ratio = 1.04, 95% CI 2-sided [0.82 to 1.32]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.5573, Negative binomial; Model includes treatment group, region, background therapy, number of exacerbations in the previous year; Rate ratio = 1.08, 95% CI 2-sided [0.84 to 1.37]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.8644, Negative binomial; Model includes treatment group, region, background therapy, number of exacerbations in the previous year; Rate ratio = 1.02, 95% CI 2-sided [0.80 to 1.30]

3. Secondary Outcome: Mean Change From Baseline to Week 56 in Pre-bronchodilator FEV1 (L) Value for Patients With Baseline EOS>=220/uL
Description: Pre-bronchodilator FEV1 (L) is collected at Weeks 0, 4, 8, 16, 24, 32, 40, 48, and 56. Baseline is the last non-missing value with quality (acceptable or borderline quality grade) prior to the first dose of study treatment.
Time Frame: First IP up to end of treatment Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 325 | 322 | 347 | 344
Liter | 0.021 (0.346) | 0.011 (0.289) | 0.033 (0.291) | 0.016 (0.292)
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Test type: Superiority; p = 0.5043, Mixed Models Analysis; Model includes treatment group, baseline FEV1 value, EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = 0.015, 95% CI 2-sided [-0.029 to 0.059]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.7691, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.007, 95% CI 2-sided [-0.051 to 0.037]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.3767, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.024 to 0.064]

4. Secondary Outcome: Mean Change From Baseline in SGRQ Total Score for Patients With Baseline EOS>=220/uL
Description: SGRQ is from 50-item PRO instrument. The SGRQ total score is expressed as a percentage of overall impairment, in which 100% means the worst possible health status and 0 indicates the best possible health status.
Time Frame: First IP up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 331 | 329 | 354 | 349
Percentage | -7.733 (14.996) | -8.674 (17.910) | -7.257 (15.989) | -6.863 (16.344)
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Test type: Superiority; p = 0.3636, Mixed Models Analysis; Model includes treatment group, baseline SGRQ score, EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = -1.011, 95% CI 2-sided [-3.192 to 1.171]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.2106, Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.388, 95% CI 2-sided [-3.562 to 0.786]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.5851, Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.602, 95% CI 2-sided [-2.763 to 1.560]

5. Secondary Outcome: Mean Change From Baseline in CAT Total Score for Patients With Baseline EOS>=220/uL
Description: CAT is an 8-item PRO developed to measure the impact of COPD on health status. The instrument uses semantic differential six-point response scales. A CAT total score is the sum of item responses. Score ranges from 0 to 40 with higher scores indicative of greater COPD impact on health status.
Time Frame: First IP up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 332 | 331 | 354 | 350
Score on a scale | -2.18 (6.78) | -2.43 (7.18) | -2.36 (6.67) | -2.36 (6.54)
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Test type: Superiority; p = 0.8525, Mixed Models Analysis; Model includes treatment group, baseline CAT total score, EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.82 to 0.99]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.9870, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.91 to 0.89]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.8204, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.00 to 0.79]

6. Secondary Outcome: Mean Change From Baseline in E-RS: COPD Total Score for Patients With Baseline EOS>=220/uL
Description: The E-RS: COPD is an 11-item PRO developed to evaluate the severity of respiratory symptoms of COPD. Summation of E-RS: COPD item responses produces a total score ranging from 0 to 40, with higher scores indicating greater severity.
Time Frame: First IP up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 316 | 302 | 317 | 325
Score on a scale | -1.657 (5.701) | -2.219 (6.381) | -1.593 (5.665) | -1.137 (5.935)
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Test type: Superiority; p = 0.2636, Mixed Models Analysis; Model includes treatment group, baseline total score, EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.102 to 0.301]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.4087, Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.296, 95% CI 2-sided [-0.998 to 0.406]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.2336, Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.425, 95% CI 2-sided [-1.125 to 0.275]

7. Secondary Outcome: Mean Change From Baseline in Total Rescue Medication Use (Number of Puffs Per Day) for Patients With Baseline EOS>=220/uL
Description: The number of rescue medication inhalations and nebulizer treatments taken are recorded by the patient in the eDiary twice daily. Total rescue medication use is the sum of daytime and night-time use.
Time Frame: First IP up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Puffs/day
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 305 | 290 | 310 | 314
Puffs/day | -0.36 (3.04) | -0.24 (3.36) | -0.17 (3.02) | 0.23 (3.55)
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Test type: Superiority; p = 0.0012, Mixed Models Analysis; Model includes treatment group, baseline rescue med. use, EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.642, 95% CI 2-sided [-1.029 to -0.254]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.0852, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.340, 95% CI 2-sided [-0.727 to 0.047]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.0650, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.364, 95% CI 2-sided [-0.750 to 0.023]

8. Secondary Outcome: Mean Change From Baseline in Proportion of Nights With Awakenings Due to Respiratory Symptoms for Patients With Baseline EOS>=220/uL
Description: Change from baseline to Week 56 in proportion of nights with awakenings due to respiratory symptoms.
Time Frame: First IP up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Proportion of nights
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 316 | 298 | 321 | 322
Proportion of nights | -0.092 (0.297) | -0.131 (0.332) | -0.084 (0.334) | -0.053 (0.345)
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Test type: Superiority; p = 0.0415, Mixed Models Analysis; Model includes treatment group, baseline prop. of nights awakens., EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.041, 95% CI 2-sided [-0.081 to -0.002]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.0069, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.055, 95% CI 2-sided [-0.094 to -0.015]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.2008, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.026, 95% CI 2-sided [-0.065 to 0.014]

9. Secondary Outcome: Number of Participants by Number of COPD Exacerbations Based on EXACT-PRO for Patients With Baseline EOS>=220/uL
Description: The EXACT-PRO is a 14-item PRO instrument developed to assess the frequency, severity and duration of COPD exacerbations. Respondents are instructed to complete the electronic diary (eDiary) each evening just prior to bedtime and to answer the questions while considering their experiences "today". The daily EXACT-PRO total score is recorded and has a range of 0-100 with higher scores indicative of greater severity. COPD exacerbation event frequency is calculated based on comparison of the baseline score with daily total scores. An increase of EXACT-PRO total score ≥9 for 3 days or ≥12 for 2 days indicates a COPD exacerbation event has occurred.
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, EOS>=220/uL
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 377 | 394 | 385 | 388
Participants
  0 | 166 | 173 | 162 | 159
  1 | 108 | 107 | 113 | 119
  2 | 45 | 51 | 56 | 46
  3 | 21 | 27 | 25 | 27
  4 | 14 | 16 | 13 | 13
  5 | 8 | 8 | 9 | 12
  6 | 7 | 6 | 4 | 7
  7 | 2 | 4 | 1 | 2
  8 | 4 | 1 | 2 | 1
  9 | 0 | 1 | 0 | 1
  10 | 2 | 0 | 0 | 0
  11 | 0 | 0 | 0 | 1

10. Secondary Outcome: Severity of EXACT-PRO for Patients With Baseline EOS>=220/uL
Description: The EXACT-PRO is a 14-item PRO instrument developed to assess the frequency, severity and duration of COPD exacerbations. Respondents are instructed to complete the electronic diary (eDiary) each evening just prior to bedtime and to answer the questions while considering their experiences "today". The daily EXACT-PRO total score has a range of 0-100 with higher scores indicative of greater severity. Severity of the study is the highest score of EXACT-PRO.
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 211 | 221 | 223 | 229
Score on a scale | 50.3 (12.30) | 52.1 (11.3) | 51.2 (11.0) | 51.0 (11.7)

11. Secondary Outcome: Duration of COPD Exacerbation Based on EXACT-PRO Score for Patients With Baseline EOS>=220/uL
Description: The EXACT-PRO is a 14-item PRO instrument developed to assess the frequency, severity and duration of COPD exacerbations. Respondents are instructed to complete the electronic diary (eDiary) each evening just prior to bedtime and to answer the questions while considering their experiences "today". The daily EXACT-PRO total score has a range of 0-100 with higher scores indicative of greater severity. COPD exacerbation event frequency is identified by comparing the baseline score with daily total scores. An increase in EXACT-PRO total score ≥9 for 3 days or ≥12 for 2 days indicate an event has occurred. Event duration is calculated after identification of the following five parameters: 1) onset; 2) three-day rolling average; 3) maximum observed value; 4) threshold for improvement; and 5) recovery. That is, duration of the exacerbation is the time elapse between onset and recovery of the event.
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 211 | 221 | 223 | 229
Days | 110.1 (114.0) | 96.1 (109.3) | 99.8 (114.8) | 99.9 (113.9)

12. Secondary Outcome: Annual EXACT-PRO Exacerbation Rate Over 56 Weeks Treatment Comparison for Patients With Baseline EOS>=220/uL
Description: The EXACT-PRO is a 14-item PRO instrument developed to assess the frequency, severity and duration of COPD exacerbations. Respondents are instructed to complete the electronic diary (eDiary) each evening just prior to bedtime and to answer the questions while considering their experiences "today". The daily EXACT-PRO total score has a range of 0-100 with higher scores indicative of greater severity. Event frequency is calculated by comparing the baseline with daily total scores. An increase in EXACT-PRO total score ≥9 for 3 days or ≥12 for 2 days indicate an event has occurred. Annual EXACT-PRO exacerbation rate is the number of exacerbations per year. Its raw rate is calculated by number of exacerbations divided by the treatment period and then normalized to an annual rate, and is estimated by negative binomial model. Rate ratio between two treatment groups is also estimated through this model.
Time Frame: Immediately following the first IP dose through week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 377 | 394 | 385 | 388
Exacerbations per year | 1.20 [1.05 to 1.37] | 1.21 [1.06 to 1.37] | 1.13 [0.99 to 1.29] | 1.23 [1.08 to 1.40]
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Test type: Superiority; p = 0.8158, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, number of exacerbations in the previous year; Rate ratio = 0.98, 95% CI 2-sided [0.81 to 1.18]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.8378, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, number of exacerbations in the previous year; Rate ratio = 0.98, 95% CI 2-sided [0.82 to 1.18]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.3759, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, number of exacerbations in the previous year; Rate ratio = 0.92, 95% CI 2-sided [0.76 to 1.11]

13. Secondary Outcome: Number of Participants Having at Least 1 COPD Exacerbation for Patients With Baseline EOS>=220/uL
Description: A COPD exacerbation is defined by symptomatic worsening COPD requiring systemic corticosteroids, antibiotics, or an inpatient hospitalization/death due to COPD.
Time Frame: Immediately following first IP dose up to week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 377 | 394 | 386 | 388
Participants | 203 | 241 | 214 | 208
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Proportion of participants with >=1 COPD exacerbation; Test type: Superiority; p = 0.9141, Cochran-Mantel-Haenszel; CMH test controlling for EOS cohort, region, and background therapy; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.76 to 1.36]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Proportion of participants with >=1 COPD exacerbation; Test type: Superiority; p = 0.0323, Cochran-Mantel-Haenszel; CMH test controlling for EOS cohort, region, and background therapy; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.03 to 1.87]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Proportion of participants with >=1 COPD exacerbation; Test type: Superiority; p = 0.5109, Cochran-Mantel-Haenszel; CMH test controlling for EOS cohort, region, and background therapy; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.82 to 1.48]

14. Secondary Outcome: Time to First COPD Exacerbation
Description: Time to first COPD exacerbation is from the randomization date to the first occurrence of COPD exacerbation.
Time Frame: Immediately following IP dose to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 377 | 394 | 386 | 388
Days | 315 [244 to 380] | 260 [225 to 291] | 322 [278 to 373] | 337 [261 to 400]

15. Secondary Outcome: Annual COPD Exacerbation Rate Associated With ER or Hospitalization Over 56 Weeks Treatment Comparison for Patients With Baseline EOS>=220/uL
Description: Annual COPD exacerbations rate that result in ER or hospitalization is calculated by number of exacerbations resulting ER or hospitalization divided by the treatment period and then normalized to an annual rate, and is estimated by negative binomial model. Rate ratio between two treatment groups is also estimated through this model.
Time Frame: Immediately following the first IP dose through week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 377 | 394 | 386 | 388
Exacerbations per year | 0.22 [0.17 to 0.29] | 0.29 [0.23 to 0.36] | 0.22 [0.17 to 0.28] | 0.32 [0.26 to 0.40]
Statistical Analysis 1: Comparison: Benralizumab 10 mg vs Placebo; Test type: Superiority; p = 0.0287, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, previous year exacerbations associated with hospitalization (Y/N); Rate ratio = 0.68, 95% CI 2-sided [0.49 to 0.96]
Statistical Analysis 2: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.4631, Negative binomial; [statistical method as in outcome 15, analysis 1]; Rate ratio = 0.89, 95% CI 2-sided [0.65 to 1.22]
Statistical Analysis 3: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.0185, Negative binomial; [statistical method as in outcome 15, analysis 1]; Rate ratio = 0.67, 95% CI 2-sided [0.48 to 0.94]

16. Secondary Outcome: Number of Participants Had COPD-related Healthcare Encounter for Patient With Baseline EOS>=220/uL
Description: Types of healthcare encounter: Hospitalisations (inc. intensive care and/or general care), Emergency department visits, Unscheduled outpatients visits, Home visits, Telephone calls, and ambulance transports.
Time Frame: Immediately following first IP dose up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 377 | 394 | 386 | 388
Participants
  Hospitalisations | 45 | 67 | 48 | 59
  Emergency department | 49 | 72 | 58 | 71
  Unscheduled outpatient visits | 208 | 230 | 225 | 211
  Home visits | 14 | 20 | 17 | 14
  Telephone calls | 98 | 112 | 109 | 114
  Ambulance transports | 10 | 19 | 20 | 22

17. Secondary Outcome: Duration of Study Treatment Administration
Description: Duration of study treatment is calculated from first dose date to last dose date + 1 day.
Time Frame: From first dose date to last dose date, 48 weeks per protocol.
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 561 | 563 | 562 | 568
Days | 307.4 (80.38) | 302.2 (84.62) | 303.0 (88.48) | 308.8 (78.95)

18. Secondary Outcome: Serum Concentration of Benralizumab
Description: PK serum samples were collected pre-dose at each visit.
Time Frame: Pre-first dose and pre-dose at end of treatment (week 56).
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg
Number analyzed (Participants) | 558 | 560 | 552
ng/mL
  Baseline: number analyzed (Participants) | 555 | 559 | 548
  Baseline | NA (NA) — <LLOQ (Lower limit of quantification) | NA (NA) — <LLOQ (Lower limit of quantification) | NA (51.95) — <LLOQ (Lower limit of quantification)
  Week 56: number analyzed (Participants) | 399 | 370 | 384
  Week 56 | 42.51 (384.81) | 222.92 (248.24) | 594.33 (321.66)

19. Secondary Outcome: Immunogenicity of Benralizumab
Description: Anti-drug antibody (ADA) responses such as ADA prevalence, ADA incidence, ADA persistently positive counts, etc. were presented.
Time Frame: Pre-treatment until end of follow-up, week 60 per protocol.
Population: Safety analysis set. For each parameter, the number of subjects at risk is to be analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 10 mg | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 561 | 563 | 562 | 568
Participants
  ADA prevalence | 70 | 52 | 77 | 26
  ADA incidence: number analyzed (Participants) | 554 | 554 | 542 | 555
  ADA incidence | 60 | 39 | 65 | 16
  Both base/post-baseline positive: number analyzed (Participants) | 554 | 554 | 542 | 555
  Both base/post-baseline positive | 9 | 8 | 5 | 10
  Only post baseline: number analyzed (Participants) | 556 | 556 | 547 | 561
  Only post baseline | 57 | 38 | 64 | 14
  Only baseline: number analyzed (Participants) | 559 | 561 | 557 | 562
  Only baseline | 4 | 6 | 8 | 2
  ADA persistently positive: number analyzed (Participants) | 554 | 554 | 542 | 555
  ADA persistently positive | 42 | 30 | 43 | 6
  ADA transiently positive: number analyzed (Participants) | 554 | 554 | 542 | 555
  ADA transiently positive | 15 | 8 | 21 | 8
  nAb prevalence | 55 | 37 | 59 | 13
  nAb incidence: number analyzed (Participants) | 554 | 554 | 542 | 555
  nAb incidence | 50 | 33 | 52 | 9

ADVERSE EVENTS:
Time Frame: From the time patient signed informed consent throughout the treatment period to the follow-up visit (week 60).
Description: Adverse events are presented according to the actual treatment the participants received. One participant randomized to Benra 10 mg was treated with Benra 30 mg, thus this participant is counted in Benra 30 mg group, and hence one less participant in Benra 10 mg, compared with patient flow summary (where participants are summarized per randomized treatment group).
Groups:
- Benra 10 mg; Benra 30 mg; Benra 100 mg; Placebo: Every 8 weeks administered subcutaneously
Arm/Group | Benra 10 mg | Benra 30 mg | Benra 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 17/561 | 21/563 | 17/562 | 19/568
Serious Adverse Events (participants affected / at risk) | 144/561 | 177/563 | 127/562 | 158/568
Other Adverse Events (participants affected / at risk) | 251/561 | 233/563 | 238/562 | 260/568
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 10 mg (N=561) | Benra 30 mg (N=563) | Benra 100 mg (N=562) | Placebo (N=568)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 7 (7) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (3) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (3)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 2 (3) | 4 (5) | 4 (4)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal artery embolism (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 3 (3)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intestinal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 19 (20) | 22 (25) | 9 (10) | 30 (34)
Pneumonia bacterial (Infections and infestations) | 5 (5) | 5 (7) | 2 (2) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (4) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
False positive tuberculosis test (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 1 (3) | 2 (2)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 0 (0) | 2 (2) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 4 (4) | 5 (5)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 92 (129) | 107 (136) | 80 (106) | 89 (140)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 3 (3) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penetrating aortic ulcer (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 10 mg (N=561) | Benra 30 mg (N=563) | Benra 100 mg (N=562) | Placebo (N=568)
Oedema peripheral (General disorders) | 15 (17) | 9 (9) | 17 (18) | 9 (10)
Bronchitis (Infections and infestations) | 66 (94) | 70 (100) | 63 (87) | 66 (88)
Influenza (Infections and infestations) | 11 (11) | 20 (22) | 15 (15) | 11 (12)
Lower respiratory tract infection (Infections and infestations) | 26 (27) | 22 (29) | 15 (16) | 21 (27)
Oral candidiasis (Infections and infestations) | 21 (25) | 12 (13) | 15 (20) | 12 (17)
Sinusitis (Infections and infestations) | 15 (18) | 13 (19) | 15 (21) | 20 (24)
Upper respiratory tract infection (Infections and infestations) | 68 (109) | 71 (98) | 67 (92) | 65 (89)
Urinary tract infection (Infections and infestations) | 24 (34) | 24 (26) | 28 (32) | 18 (22)
Viral upper respiratory tract infection (Infections and infestations) | 61 (73) | 47 (68) | 60 (92) | 70 (93)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 12 (12) | 17 (20) | 15 (15)
Headache (Nervous system disorders) | 19 (20) | 16 (17) | 27 (34) | 24 (36)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 10 (13) | 20 (24) | 24 (34)
Hypertension (Vascular disorders) | 17 (22) | 16 (17) | 12 (12) | 21 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2015-07-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT02155660/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT02155660/SAP_001.pdf